CLINICAL TRIAL: NCT03149640
Title: Double-blinded Multicenter Randomized Controlled Trial Comparing Inhaled Amikacin Versus Placebo to Prevent Ventilator Associated Pneumonia
Brief Title: Study Comparing Inhaled Amikacin Versus Placebo to Prevent Ventilator Associated Pneumonia
Acronym: AMIKINHAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PHRN15-SE / AMIKINHAL
Record Dates: First submitted 2017-05-02; First posted 2017-05-11 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2022-11

CONDITIONS: Pneumonia, Ventilator-Associated
Keywords: Prevention; inhaled amikacin; placebo
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhaled amikacin (Experimental): Inhaled amikacin at day 4, day 5 and day 6 of invasive mechanical ventilation: 20 mg/kg of ideal body weight, maximum 2 g per day.
  Interventions: Drug: Inhaled amikacin
- Placebo (Placebo Comparator): Once a day, inhaled placebo at day 4, day 5 and day 6 of invasive mechanical ventilation.
  Interventions: Drug: Inhaled placebo

INTERVENTIONS:
Drug: Inhaled amikacin — Once a day, inhaled amikacin at day 4, day 5 and day 6 of invasive mechanical ventilation: 20 mg/kg of ideal body weight, maximum 2 g per day.
  Arms: Inhaled amikacin
Drug: Inhaled placebo — Once a day, inhaled placebo at day 4, day 5 and day 6 of invasive mechanical ventilation.
  Arms: Placebo

SUMMARY:
The objective of the study is to prove that after the third day of invasive mechanical ventilation a three-day course of inhaled amikacin reduces the incidence of subsequent VAP.

Parallel two group double blind randomized controlled clinical trial. Individual randomization, performed on day 4 of invasive mechanical ventilation, will be stratified on centre in order to account for variations in VAP prevention bundle implementation and use of systemic antibiotics the day of randomization. Patients will be treated three consecutive days with inhaled amikacin or placebo. Patients will be followed up daily in the intensive care unit for the occurrence of VAP according to international guidelines until day 28.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years the day of inclusion
* Mechanical ventilation through an endotracheal tube for more than three consecutive days (72h)
* Written informed consent of the patient or a proxy
* Patients covered by or having the rights to French social security
* Negative pregnancy test, at the time of inclusion, in women of childbearing potential

Exclusion Criteria:

* Suspicion or confirmed VAP the day of inclusion
* Clinical indication for systemic aminoglycoside therapy the day of inclusion : as deemed necessary by the clinician in charge
* Stage 2 or 3 KDIGO* classification acute kidney injury the day of inclusion excepted in patients undergoing renal replacement therapy
* Chronic kidney failure : baseline glomerular filtration lower than 30 mL/min
* Patient scheduled for extubation within the next 24h
* Patient ventilated through an endotracheal tube for more than four consecutive days before inclusion (96h)
* Patient ventilated through a tracheostomy
* Patients allergic to aminoglycosides
* Myasthenia gravis
* Known pregnant women at the time of inclusion and lactating patients
* Known guardianship or trusteeship at the time of inclusion
* Patients previously included in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-06-17 (Actual)

PRIMARY OUTCOMES:
Incidence of a first VAP episode from randomization to day 28 | Patients will be followed from randomization to day 28

SECONDARY OUTCOMES:
Incidence of a first VAP episode in the subgroups of patients with tracheobronchial colonization or tracheobronchitis | At randomization
Incidence of VAP due to Gram negative amikacin sensitive bacteria | Patients will be followed from randomization to day 28
Clinical pulmonary infection score evolution | Patients will be followed from randomization to day 28
Ventilator associated events incidence | Patients will be followed from randomization to day 28
Number of systemic antibiotics administered per day | Patients will be followed from randomization to day 28
Number of days with at least one administration of a systemic antibiotic | Patients will be followed from randomization to day 28
Incidence of antibiotic resistant bacteria isolated on clinical and hygiene samples | Patients will be followed from randomization to day 28
Incidence of acute kidney injury | Patients will be followed from randomization to day 28
Days spent on mechanical ventilation from randomization to day 90 | Patients will be followed from randomization to day 90
Days from randomization to the first successful spontaneous breathing trial | Days from randomization to day 90 max
Days spent in the intensive care unit and in the hospital | Patients will be followed from randomization to discharge (day 90 max)
Day 90 mortality | Day 90
Incidence of bacteria producing extended spectrum beta-lactamase or high level derepressed celphalosporinase, of vancomycin resistant Enterococcus Sp. on rectal samples | Day 28
Relative bacterial species composition of respiratory and digestive microbiota | Patients will be followed from randomization to day 28
Maximum serum Concentration | Between Hour 0-Hour 8, between Hour 8-Hour 16 and between Hour 16-Hour 24
Maximum sputum Concentration | Between Hour 0-Hour 8, between Hour 8-Hour 16 and between Hour 16-Hour 24
Area Under the Curve | Between Hour 0-Hour 8, between Hour 8-Hour 16 and between Hour 16-Hour 24
To evaluate the effects on respiratory mechanics of nebulization of amikacin by evaluating the benefit balance / risk | Measurements at 8 hours, 12 hours and 24 hours after the end of nebulization
  benefit : Improvement of respiratory mechanics by pharmacological effect risk : Degradation of respiratory mechanics by bronchospastic secondary effect, drug deposition in the intubation probe

CONTACTS AND LOCATIONS:
Overall Officials: Stephan EHRMANN, MD-PhD, Principal Investigator — University Hospital, Tours
Locations (18):
- France (18):
  - Service de Réanimation Chirurgicale, Angers
  - Service de Réanimation Médicale - CH d'Angoulême, Angoulême
  - Service de Réanimation Polyvalente, Argenteuil
  - Service de Réanimation Médicale - Hôpital Louis Mourier, Colombes
  - Service de Réanimation, Dijon
  - Service de Réanimation Médicale - CHD Les Oudairies, La Roche-sur-Yon
  - Service de Réanimation, Le Mans
  - Service de Réanimation Médicale - Hôpital La Croix-Rousse, Lyon
  - Service de Réanimation Médicale, Orléans
  - Service de Réanimation Médicale - Hôpital Pitié Salpêtrière, Paris
  - Service de Réanimation Médicale - CHU La Milétrie, Poitiers
  - Service de Réanimation Médicale, Poitiers
  - Service de Réanimation Médicale - CHU Pontchaillou, Rennes
  - Service de Réanimation Médicale - CHU Rouen, Rouen
  - Service de Réanimation Médicale - Hôpital Charles Nicolle, Rouen
  - Service de Réanimation - NHC, Strasbourg
  - Service de Réanimation Médicale - Hôpital de Hautepierre, Strasbourg
  - Service de Réanimation médicale, Hôpital Trousseau, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tavernier E, Barbier F, Meziani F, Quenot JP, Herbrecht JE, Landais M, Roux D, Seguin P, Schnell D, Veinstein A, Veber B, Lasocki S, Lu Q, Beduneau G, Ferrandiere M, Dahyot-Fizelier C, Plantefeve G, Nay MA, Merdji H, Andreu P, Vecellio L, Muller G, Cabrera M, Le Pennec D, Respaud R, Lanotte P, Gregoire N, Leclerc M, Helms J, Boulain T, Lacherade JC, Ehrmann S; REVA network and the CRICS-TRIGGESEP F-CRIN network. Inhaled amikacin versus placebo to prevent ventilator-associated pneumonia: the AMIKINHAL double-blind multicentre randomised controlled trial protocol. BMJ Open. 2021 Sep 14;11(9):e048591. doi: 10.1136/bmjopen-2020-048591. PMID 34521664
- [Derived] Ehrmann S, Barbier F, Demiselle J, Quenot JP, Herbrecht JE, Roux D, Lacherade JC, Landais M, Seguin P, Schnell D, Veinstein A, Gouin P, Lasocki S, Lu Q, Beduneau G, Ferrandiere M, Plantefeve G, Dahyot-Fizelier C, Chebib N, Mercier E, Heuze-Vourc'h N, Respaud R, Gregoire N, Garot D, Nay MA, Meziani F, Andreu P, Clere-Jehl R, Zucman N, Azais MA, Saint-Martin M, Gandonniere CS, Benzekri D, Merdji H, Tavernier E; Reva and CRICS-TRIGGERSEP F-CRIN Research Networks. Inhaled Amikacin to Prevent Ventilator-Associated Pneumonia. N Engl J Med. 2023 Nov 30;389(22):2052-2062. doi: 10.1056/NEJMoa2310307. Epub 2023 Oct 25. PMID 37888914